CLINICAL TRIAL: NCT05577429
Title: The Potential of a Low Oxygen Environmental Chamber as an Aid to Exercise Training to Improve Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: National Sports Institute of Malaysia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 20225950-9155; ISNRG003/2020 (Other Grant/Funding Number: National Sports Institute of Malaysia)
Record Dates: First submitted 2022-09-29; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Overweight; Physical Inactivity; Healthy
Keywords: Hypoxia; Overweight; Glucose tolerance; Exercise
MeSH Terms: conditions — Overweight; Sedentary Behavior; Hypoxia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be required to complete 3 exercise interventions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity exercise under normoxia (Placebo Comparator): The participants will perform low-moderate intensity cycling exercise at 90% lactate threshold (LT) (determined during LT test) under normoxia (FiO2: 20.9%) for 60 minutes on a cycle ergometer. Immediately after exercise oral glucose tolerance test (OGTT) will be determined with 24-hour glucose concentration will be monitored continuously. Circulatory factors will be determined pre, immediately after exercise and 24 hours after exercise.
  Interventions: Other: Low-moderate intensity exercise under normoxia
- Moderate intensity exercise under hypoxia (Experimental): The participants will perform low-moderate intensity cycling exercise at 90% lactate threshold (LT) (determined during LT test) under hypoxia (FiO2: 16.5-14.8%) for 60 minutes on a cycle ergometer. Immediately after exercise oral glucose tolerance test (OGTT) will be determined with 24-hour glucose concentration will be monitored continuously. Circulatory factors will be determined pre, immediately after exercise and 24 hours after exercise.
  Interventions: Other: Low-moderate intensity exercise under moderate hypoxia; Other: Low-moderate intensity exercise under high hypoxia

INTERVENTIONS:
Other: Low-moderate intensity exercise under normoxia — The participant will perform the exercise interventions consisting of cycling at the 90% lactate threshold at normoxia (fraction oxygen: 20.9%) for 60 minutes on separate days (5-7 days). Immediately after exercise oral glucose tolerance test (OGTT) and 24-hour glucose concentration will be monitored continuously. Pre, post and post-24 h circulatory markers will be determined.
  Arms: Moderate intensity exercise under normoxia
Other: Low-moderate intensity exercise under moderate hypoxia — The participant will perform the exercise interventions consisting of cycling at the 90% lactate threshold at normoxia (fraction oxygen: 16.5%) for 60 minutes on separate days (5-7 days). Immediately after exercise oral glucose tolerance test (OGTT) and 24-hour glucose concentration will be monitored continuously. Pre, post and post-24 h circulatory markers will be determined.
  Arms: Moderate intensity exercise under hypoxia
Other: Low-moderate intensity exercise under high hypoxia — The participant will perform the exercise interventions consisting of cycling at the 90% lactate threshold at normoxia (fraction oxygen: 14.8%) for 60 minutes on separate days (5-7 days). Immediately after exercise oral glucose tolerance test (OGTT) and 24-hour glucose concentration will be monitored continuously. Pre, post and post-24 h circulatory markers will be determined.
  Arms: Moderate intensity exercise under hypoxia

SUMMARY:
Obesity is a major global health issue and a primary risk factor for metabolic-related disorders. While physical inactivity is one of the main contributors to obesity, it is a modifiable risk factor with exercise training as an established, non-pharmacological treatment to prevent the onset of metabolic-related disorders, including obesity. Exposure to hypoxia via normobaric hypoxia (simulated altitude via reduced inspired oxygen fraction), termed hypoxic conditioning, in combination with exercise has been increasingly shown in the last decade to enhance blood glucose regulation and decrease body mass index, providing a feasible strategy to treat obesity.

Nonetheless, findings from studies investigating the potential for a hypoxic environment to augment the exercise training response and subsequent metabolic health are equivocal. Notably, there is a paucity of information regarding the optimal combination of exercise variables and hypoxic load (i.e. level of hypoxia) to enable an individualized and safe practice of exercising in a hypoxic environment.

In the present randomized, single-blind, cross-over study, the investigators will investigate the effects of single-bout of exercise under normoxia (FiO2, 20.9%), moderate (FiO2, 16.5%) and high normobaric hypoxic conditions (FiO2, 14.8%) (60-min cycling session at 90% LT) on 2h OGTT and 24h-glucose level in individuals with overweight. The investigators hypothesize that exercise in combination with hypoxia improves glucose homeostasis in individuals with overweight.

DETAILED DESCRIPTION:
In the present randomized, single-blind, cross-over study, participants will be exposed to normobaric 1) normoxia (oxygen level 20.9%), 2) moderate hypoxia (oxygen level 16.5%) and 3) high hypoxia (oxygen level 14.8%) 1) during exercise (60 minutes on a cycle ergometer) at 90% LT. Participants will be randomly assigned to each condition (computer-generated randomization plan), separated by a washout period (5-7 days). To accomplish this, participants will exercise in an environmental chamber in which oxygen concentration of the ambient air and, as such, oxygen levels can be closely controlled and monitored. Participants will cycle for 60 minutes at a 90% lactate threshold (LT), determined by an LT test.

Visit 1 (Screening and consent):

Introduction to the research team and tour of the facility. Complete and sign the Adult Pre-Exercise Screening System form. Complete and sign the consent information form.

Visit 2:

Body composition screening using bioimpedance analysis (Inbody 770, Cerritos, CA, USA) Blood pressure screening. Lactate threshold test-participants will be riding a Velotron cycle ergometer (Racermate, Seattle, USA) with an initial load of 50 Watts. The load increased progressively in 15 Watts increments every 4 minutes, with participants maintaining a constant pedal frequency (cadence ~90 rpm) until reaching LT.

Visit 3:

Baseline oral glucose tolerance test (OGTT)-Participants will be consumed 75 grams of glucose dissolved in water (Glucolin glucose powder) and blood samples will be collected to determine baseline glucose and insulin level.

Visit 4:

Attachment of Continuous Glucose Monitor (CGM) (FreeStyle Libre, Abbott Diabetes Care, Witney, UK) will be placed on the back of the upper arm as recommended by the manufacturer.

Visit 5:

Pre-exercise blood sampling-to determine plasma glucose, insulin and circulatory factors.

Participants will be 60 minutes of cycling bouts at 90% of LT under simulated altitude exposure (normoxia or two hypoxic conditions) in the environmental chamber.

Post-exercise blood sampling-2 hours OGTT will be performed immediately following each experimental trial to determine glucose homeostasis and circulatory factors.

Visit 6:

Post-exercise 24 hours blood sampling-to determine glucose homeostasis and circulatory factors.

Removal of CGM

ELIGIBILITY:
Inclusion Criteria:

* BMI is between 25-29 kg/m²
* Sedentary (physical activity <150 min/week)
* No known heart or metabolic diseases (such as Type 2 diabetes)
* Not currently taking any prescribed medication
* No reported musculoskeletal injuries recently
* Not exposed to hypoxia >1000 m prior to the study

Exclusion Criteria:

* Impaired glucose tolerance (2 hour glucose: >7.8 - 11.1 mmol/L)
* Type 2 diabetes mellitus
* Obstructive sleep apnea
* Chronic obstructive pulmonary disease

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial plasma glucose concentration | Change of fasting and postprandial plasma glucose concentrations (mmol/L) compared to moderate intensity exercise under normoxia (20.9% oxygen) at immediately after exercise (2 hour oral glucose tolerance test).
  Change of plasma glucose concentration immediately post-exercise under hypoxia (14.8-16.5% oxygen) compared to normoxia.
Fasting and postprandial plasma insulin concentration | Change of fasting and postprandial plasma insulin concentrations (mU/L) compared to moderate intensity exercise under normoxia (20.9% oxygen) at immediately after exercise (2 hour oral glucose tolerance test).
  Change of plasma insulin concentration immediately post-exercise under hypoxia (14.8-16.5% oxygen) compared to normoxia.

SECONDARY OUTCOMES:
Average 24 hours glucose concentration | Change of average glucose concentration compared to moderate intensity exercise under normoxia (20.9% oxygen) up to 24 hour after exercise.
  Glucose concentration will be measured in the interstitial fluid of the subcutaneous adipose tissue every 15 min using a glucose sensor (FreeStyle Libre, Abbott Diabetes Care, Witney, UK), which will be inserted subcutaneously, under skin on the arm, and will be connected to a continuous glucose monitor (Abbott FreeStyle Libre™). The cumulative effects of the acute single-bout exercise will be determined using the average 24 hours glucose levels collected on post 24 h.
Circulating concentration of fibroblast growth factor 21 (FGF-21) | Change of concentrations of FGF-21 compared to moderate intensity exercise under normoxia (20.9% oxygen) immediately after exercise and at 24 hours after exercise.
  Moderate intensity exercise under moderate-high hypoxia compared to normoxia. Pre, immediate post and post 24 hours blood will be sampled and analysed for circulating markers by means of ELISA
Circulating concentration of apelin | Change of concentrations of apelin compared to moderate intensity exercise under normoxia (20.9% oxygen)immediately after exercise and at 24 hours after exercise.
  Moderate intensity exercise under moderate-high hypoxia compared to normoxia. Pre, immediate post and post 24 hours blood will be sampled and analysed for circulating markers by means of ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Donny Camera, PhD, Principal Investigator — Swinburne University of Technology
Locations (1):
- National Sports Institute of Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No